CLINICAL TRIAL: NCT03010267
Title: An Open-label, Randomized, Crossover Study to Evaluate the Pharmacokinetics and Safety of a Fixed Dose Combination of Raloxifen/Cholecalciferol Compared With Coadministration of Raloxifen and Cholecalciferol in Healthy Male Subjects
Brief Title: DP-R213 Phase 1 Pharmacokinetics Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DP-CTR213-I-04
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: DP-R213
MeSH Terms: interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RT group (Experimental): combination dose of Raloxifene and Cholecaliferol and DP-R213 in order
  Interventions: Drug: DP-R213; Drug: Raloxifene; Drug: Cholecaliferol
- TR group (Experimental): combination dose of Raloxifene and Cholecaliferol and DP-R213 in order
  Interventions: Drug: DP-R213; Drug: Raloxifene; Drug: Cholecaliferol

INTERVENTIONS:
Drug: DP-R213 — Investigational product is prescribed to all of randomized subjects
Drug: Raloxifene — Investigational product is prescribed to all of randomized subjects
Drug: Cholecaliferol — Investigational product is prescribed to all of randomized subjects

SUMMARY:
A randomized, open-label, crossover, Phase I clinical trial to compare the pharmacokinetics of DP-R213 (Raloxifenel and Cholecaliferol fixed dose combinations) in comparison to each component administered alone in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* IBW ±20%
* Signed the informed consent form prior to the study participation

Exclusion Criteria:

* Clinically significant disease
* Previously donate whole blood within 2 months or component blood within 1 month
* Clinically significant allergic disease
* Taken IP in other trial within 3 months
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | up to 96 hours post dose
Peak Plasma Concentration (Cmax) | up to 96 hours post dose

REFERENCES:
- [Derived] Lee HW, Kang WY, Gwon MR, Choi EJ, Kim EH, Cho K, Lee B, Seong SJ, Yoon YR. A randomized, open-label, single-dose, two-way crossover study to assess the pharmacokinetics between two tablets of fixed-dose combination formulation with raloxifene and cholecalciferol and concomitant administration of each agents in healthy male volunteers. Transl Clin Pharmacol. 2022 Sep;30(3):136-144. doi: 10.12793/tcp.2022.30.e13. Epub 2022 Sep 15. PMID 36247744